CLINICAL TRIAL: NCT06533189
Title: Developing a Whole-body Magnetic Resonance Imaging and Diffusion-weighted Imaging State-of-the-art Protocol, a Pilot Study
Brief Title: Developing a Whole-body MRI and Diffusion-weighted Imaging State-of-the-art Protocol: a Pilot Study
Acronym: WANDA
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 6171
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Whole Body Imaging; Cancer; Genetic Predisposition
Keywords: MRI; Whole Body MRI; Genetic Predisposition to Cancer
MeSH Terms: conditions — Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Enhanced Diffusion Software — Application of specific sequences with the use of Enhanced Diffusion Software during Patient MRI

SUMMARY:
Whole-body magnetic resonance imaging (WB-MRI) is a non-ionizing imaging method that can provide WB coverage using essential imaging contrasts with the possibility to include sequences focusing in specific body-regions as needed per case. WB-MRI is increasingly being used for the management of cancer patients, especially metastatic ones. An integral part of WB-MRI is becoming whole-body diffusion-weighted MRI (WB-DWI) which is a non-invasive tool used for staging and response evaluation in oncologic practice. WB-DWI is an inherently noisy technique, resulting in it accounting for more than 50% of the acquisition time of conventional whole-body MRI studies with overall duration at least 1-hour. Reducing acquisition times, without compromising image or diagnostic quality would facilitate the wider adoption of clinical WBDWI, reducing costs, and improving the patient experience

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Patients with diagnosis of multiple myeloma, lymphoma, lung, prostate, breast, colorectal and gynecologic cancers;
* Patients with genetic syndromes responsible for an increased predisposition to neoplasms (e.g. Li Fraumeni syndrome);
* Signed written informed consent to personal data treatment for research purposes

Exclusion Criteria:

* Age <18 years old;
* Refusal to sign the written informed consent to personal data treatment for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncologic patients (with multiple myeloma, lymphoma, melanoma and metastatic cancer, such as prostate, breast and gynecologic cancers. Another application of WB-MRI is the imaging of patients with certain cancer predisposition syndromes
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Radiologists' satisfaction of the quality of images | 18 months
  Radiologists' satisfaction of the quality of images after applying noise reduction methods, in terms of mean overall response rate ≥4 at the questionnaires' items

SECONDARY OUTCOMES:
Diagnostic accuracy of the de-noised WB-MRI in detecting lesions | 18 months
  Comparison of diagnostic accuracy for lesion detection after applying noise reduction methods with that of standard reference imaging modalities,
Diagnostic accuracy of the de-noised WB-MRI in detecting staging metastatic oncologic patients. | 18 months
  Comparison of diagnostic accuracy for staging neoplasms according to the reference staging system with that of standard reference imaging modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Evis Sala, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Radiologia, Roma
  - Advanced Radiology Center, Rome

IPD SHARING:
Plan to Share IPD: No